CLINICAL TRIAL: NCT06344663
Title: The Effect of Motivational Interviews to Mothers With Insufficient Milk Perception on Breastfeeding Motivation and Cortisol Level
Brief Title: Motivational Interviewing Inadequate Milk and Cortisol
Status: Recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, doctor lecturer, Kahramanmaras Sutcu Imam University
Other Study IDs: KSIU-SBF-ES-02
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Motivation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Mothers who will be included in the control group will be interviewed twice in total. Pretest data will be obtained by applying the "Personal Information Form", "Insufficient Milk Perception Scale" and "Breastfeeding Motivation Scale" during the first interview. A sample of the mothers' saliva will be taken to measure cortisol values. Four weeks after the pre-test data are obtained, post-test data will be obtained by applying the "Insufficient Milk Perception Scale" and "Breastfeeding Motivation Scale". Finally, a saliva sample will be taken to check the cortisol value again.
- intervention group: Before starting the motivational interviews, pre-test data will be obtained by applying the "Personal Information Form", "Insufficient Milk Perception Scale" and "Breastfeeding Motivation Scale" to the mothers in the intervention group. Afterwards, a sample of the mothers' saliva will be taken to measure their cortisol levels. A total of 4 sessions of motivational interviews will be held for infertile women, 1 session per week for four weeks. At the end of four weeks, post-test data will be obtained by applying the "Insufficient Milk Perception Scale" and "Breastfeeding Motivation Scale". A sample of the mothers' saliva will be taken to measure cortisol levels again.
  Interventions: Other: motivational interview

INTERVENTIONS:
Other: motivational interview — Before starting the interview, mothers will be informed about the interview intervals, duration, how many times it will be held, and that, unlike other interviews, the topic will be determined and the mother's opinions on this subject will be obtained. Each meeting will last approximately 15-30 minutes
  Groups: intervention group

SUMMARY:
Motivational interviewing is a technique used in many fields. No study has been found in national and international databases investigating the effect of motivational interviewing on the perception of insufficient milk, breastfeeding motivation and cortisol level. The study aimed to evaluate the effect of motivational interviews on the perception of insufficient milk, breastfeeding motivation and cortisol level.

DETAILED DESCRIPTION:
Motivational interviewing; It is an evidence-based and client-centered approach that finds and eliminates the person's complex emotions, motivates, and increases the person's self-efficacy and motivation in the decision-making process. Breast milk is the only physiological baby food that contains the nutrients necessary for babies' absorption in appropriate quantity and quality. It is very important for the mother and baby's health that the mother starts breastfeeding her baby as early as possible and that the baby is fed only breast milk for the first six months. The perception of insufficient milk is defined as the mother thinking that she cannot produce milk or believing that there is too little milk in her breasts. The main reasons are; The mother's stay in the hospital longer than normal during the postpartum period, the mother's separation from her baby, and therefore the late establishment of the emotional bond between the mother and the baby may trigger the perception of insufficient milk. Cortisol is a glucocorticoid steroid hormone that is released in the human body during stress and whose release is regulated through the hypothalamic-pituitary adrenal (HPA) system. Stress and fear of birth cause insufficient milk secretion. Stress and fear in the mother can prevent early skin-to-skin contact between the mother and the baby by affecting the oxytocin hormone.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 and over
* Those who feed their babies only with breast milk
* Do you believe that you produce enough milk to feed your baby?" in the Insufficient Milk Perception Scale. Those who answered "No" to the question
* Having given birth at 37>gestational weeks
* Having a baby weighing at least 2500 grams
* Giving birth vaginally
* Primiparous

Exclusion Criteria:

* Cannot speak Turkish
* Mothers who did not agree to participate in the research

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers with the perception of insufficient milk
Study Population: Mothers with the perception of insufficient milk
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Insufficient Milk Perception Scale (ANN) | 1 month
  The Insufficient Milk Perception Scale is a scale developed by McCarterSpaulding (2001) to measure mothers' beliefs about whether they produce sufficient milk. It consists of 6 questions. A minimum score of 0 and a maximum score of 50 can be obtained from this scale. A high score indicates that the mother's perception of adequate milk is high

SECONDARY OUTCOMES:
Breastfeeding Motivation Scale (EMS) | 1 month
  Based on the self-determination theory of the "Breastfeeding Motivation Scale" (EMS), Peleg et al. It was developed by in 2015. After the scale was applied to the sample group, factor analysis was performed and it was determined that it had 5 factors. These factors; It consists of integrated, identified, introjected, external regulation and internal motivation. No total score is obtained from the scale. As the score obtained from the sub-dimension of the scale increases, the motivation representing that sub-dimension also increases

OTHER OUTCOMES:
Visual Analog Scale (VAS) | 1 month
  Satisfaction Level Rating with Motivational Interviewing Application is a scale developed by Hayes and Patterson in 1921, used to express some values that cannot be measured with numbers. In the satisfaction rating scale, which was created by taking the Visual Analog Scale as an example, the mother's satisfaction level will be marked on this line by writing "not at all satisfied" on one end and "very satisfied" on the other end.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Karataş Okyay, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Eda Sever, Kahramanmaraş, Onikişubat, Turkey (Türkiye)